CLINICAL TRIAL: NCT02354794
Title: Effect of Oral Supplementation With One Form of L-arginine on Vascular Endothelial Function in Healthy Subjects Featuring Risk Factors Related to the Metabolic Syndrome.
Brief Title: Effect of Arginine Supplementation in the Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: Institut de Recherche Pierre Fabre (Other); Hospital Avicenne (Other); Adeprina (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, PU-PH in University Hospitals Paris-Seine-Saint-Denis-APHP-University Hospital Avicenne / Jean Verdier, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: FRMA13-1; 2013-A01043-42 (Other: ANSM)
Record Dates: First submitted 2014-09-24; First posted 2015-02-03 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-01

CONDITIONS: Overweight; Hypertriglyceridemic Waist
Keywords: arginine; supplementation; metabolic syndrome; endothelial function
MeSH Terms: conditions — Overweight; Hypertriglyceridemic Waist; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy subjects with 'hypertriglyceridemic waist' (Experimental): Subjects with overweight, elevated waist circumference and elevated fasting triglyceridemia.
  Intervention: see below
  Interventions: Dietary Supplement: One form of arginine; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: One form of arginine — 3 capsules containing 0.5g of one form of L-arginine (1.5g) 3 times daily (4.5g per day) for 1 month
Dietary Supplement: placebo — 3 capsules containing 0.5g cellulose (non active product) 3 times daily (4.5g per day) for 1 month

SUMMARY:
The purpose of this study is to determine whether oral supplementation with one form of arginine improves vascular endothelial function in healthy subjects with risk factors associated with the metabolic syndrome

DETAILED DESCRIPTION:
The study is a randomized crossover study including 32 subjects with risk factors associated with metabolic syndrome. In a cross-over design, each subject received oral arginine and placebo, in a randomized order, and were studied the day preceding the first day of administration of arginine (or placebo) and after 4 weeks of arginine (or placebo) supplementation. The two periods of supplementation were separated by a washout period of at least 4 weeks.

The subject were studied in the morning (when before supplementation) and in a whole day (when after supplementation).

The mornings cessions consisted of fasting blood draw and vascular explorations, including a measurement of endothelium-dependent brachial artery reactivity ("Flow mediated dilation"), directly coupled to a measurement of post-ischemic digital reactivity (with the Endo-PAT method), completed by a measurement of non-endothelium-dependent brachial artery reactivity. An analysis of the pulse wave geometry was also performed.

The whole-day cession consisted of the same fasting vascular explorations. Blood tests were performed fasting and repeated 2, 4 and 6 h after ingestion of a high-fat meal (900 kcal). Measurements of Flow mediated dilation was repeated 4h and postischemic digital reactivity were repeated 2, 4 and 6 h after ingestion of the high fat meal.

ELIGIBILITY:
Inclusion Criteria :

* Age between 18 to 60 years old
* Overweight (BMI between 25 and 30 kg/m²)
* 'Hypertriglyceridemic waist' (waist circumference > 94cm for men or > 88cm for women and fasting triglyceride levels > 150 mg/dL)

Exclusion Criteria :

* Obesity (BMI> 30 kg / m²)
* Cardiac or vascular diseases
* Diabetes
* Thyroid disease
* Systolic blood pressure > 150 mmHg or diastolic blood pressure > 90 mmHg
* Tobacco consumption > 6 cigarettes per week
* Alcohol consumption> 2 drinks per day
* Any medication (except contraceptive treatment) or dietary supplement intake that could not be arrested more than a week before the first visit for the duration of the study.
* Persons under guardianship
* Positive Hepatitis B virus (HBV), Hepatitis C virus (HCV) and HIV
* Hemoglobin < 14 g/dl (for men) or <12 g / dl (for women)
* Participation in a clinical trial within 6 months preceding the study
* Pregnant and lactating women
* For women, menstrual cycle with a duration different from 28 (± 1) days (the cycle is not controlled by a contraceptive treatment at 28 days, or he does not appear spontaneously with regularity)
* Subjects with allergies to final product components
* Contraindications to arginine intake, namely asthmatics subjects, people prone to herpes, patients with liver cirrhosis and renal failure
* Hypotensive patients for whom the use of nitroglycerin is contraindicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Physiological assessment of endothelial function in postprandial and fasting (Endothelial function was assessed by flow-mediated dilation (FMD) and peripheral arterial tonometry (EndoPAT) | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Endothelial function was assessed by flow-mediated dilation (FMD) and peripheral arterial tonometry (EndoPAT).
  FMD technique was used during the fasting test. The RHI measurements were performed the morning fasting and 2, 4, and 6 hours after administration of the high-fat meal, in the case of exploration days after supplementation. In terms of the 4h measurement, it was coupled to a FMD assessment.
  FMD was calculated as the percentage change in artery diameter at peak dilation compared with baseline and is reported as a percentage.
  The Reactive Hyperemia Index (RHI) was calculated as the ratio of the average pulse wave amplitude during hyperemia (60 to 120 s of the postocclusion period) to the average pulse wave amplitude during baseline in the occluded hand divided by the same values in the control hand and then multiplied by a baseline correction factor.
Evaluation of plasma vascular cell adhesion molecule-1 (VCAM-1) of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations of VCAM-1 will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma intercellular adhesion molecule (ICAM-1) of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations of ICAM-1 will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma E-Selectin of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations E-Selectin will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma P-Selectin of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations P-Selectin will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma Plasminogen activator inhibitor-1 (PAI-1) of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations of PAI-1) will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma C-reactive protein (CRP) of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations of CRP will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.
Evaluation of plasma Endothelin-1 of endothelial function in postprandial and fasting | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting plasma concentrations of Endothelin-1 will be determined using two custom mixed assay kits with antibody-coated beads using the Luminex xMAP technology platform for multiplexing of immunochemical bioassays.

SECONDARY OUTCOMES:
Asymmetric Dimethyl-L-Arginine (ADMA) measurement | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  - Fasting ADMA concentrations were measured by an enzyme-linked immunosorbent assay.
Amino acids measurement | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting amino acids contents was assayed by High-performance liquid chromatography (HPLC).
Nitrite measurement | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting nitrite were analyzed by Gas chromatography-mass spectrometry (GC-MS).
Complete blood count (CBC) analysis | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting and postprandial complete blood count (CBC) (was assayed using "classical clinical biochemical analyzers".
Insulin and glucose measurement | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  The fasting insulin and the fasting and postprandial glucose were assayed using "classical clinical biochemical analyzers".
Lipid profile analysis | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  - The fasting lipid profile (triglycerides, total cholesterol, HDL-cholesterol, LDL-cholesterol) and the postprandial evolution of triglycerides were measured and were assayed using "classical clinical biochemical analyzers".
Metabolomic analysis | Before the supplementation at day 0 and after the supplementation (1month after) at day 29 for each treatment
  Fasting metabolomic analysis with metabolomic approaches

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, Principal Investigator — Hospital Avicenne; François Mariotti, PhD, Study Director — AgroParisTech
Locations (1):
- Centre de Recherche sur Volontaires (CRV), Hospital Avicenne, Bobigny, Île-de-France Region, France

REFERENCES:
- [Background] Abdelhamed AI, Reis SE, Sane DC, Brosnihan KB, Preli RB, Herrington DM. No effect of an L-arginine-enriched medical food (HeartBars) on endothelial function and platelet aggregation in subjects with hypercholesterolemia. Am Heart J. 2003 Mar;145(3):E15. doi: 10.1067/mhj.2003.160. PMID 12660684
- [Background] Adams MR, Forsyth CJ, Jessup W, Robinson J, Celermajer DS. Oral L-arginine inhibits platelet aggregation but does not enhance endothelium-dependent dilation in healthy young men. J Am Coll Cardiol. 1995 Oct;26(4):1054-61. doi: 10.1016/0735-1097(95)00257-9. PMID 7560599
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Arsenault BJ, Lemieux I, Despres JP, Wareham NJ, Kastelein JJ, Khaw KT, Boekholdt SM. The hypertriglyceridemic-waist phenotype and the risk of coronary artery disease: results from the EPIC-Norfolk prospective population study. CMAJ. 2010 Sep 21;182(13):1427-32. doi: 10.1503/cmaj.091276. Epub 2010 Jul 19. PMID 20643837
- [Background] Bai Y, Sun L, Yang T, Sun K, Chen J, Hui R. Increase in fasting vascular endothelial function after short-term oral L-arginine is effective when baseline flow-mediated dilation is low: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2009 Jan;89(1):77-84. doi: 10.3945/ajcn.2008.26544. Epub 2008 Dec 3. PMID 19056561
- [Background] Balkau B, Vernay M, Mhamdi L, Novak M, Arondel D, Vol S, Tichet J, Eschwege E; D.E.S.I.R. Study Group. The incidence and persistence of the NCEP (National Cholesterol Education Program) metabolic syndrome. The French D.E.S.I.R. study. Diabetes Metab. 2003 Nov;29(5):526-32. doi: 10.1016/s1262-3636(07)70067-8. PMID 14631330
- [Background] Barringer TA, Hatcher L, Sasser HC. Potential benefits on impairment of endothelial function after a high-fat meal of 4 weeks of flavonoid supplementation. Evid Based Complement Alternat Med. 2011;2011:796958. doi: 10.1093/ecam/nen048. Epub 2011 Jun 5. PMID 18955351
- [Background] Beaumier L, Castillo L, Ajami AM, Young VR. Urea cycle intermediate kinetics and nitrate excretion at normal and "therapeutic" intakes of arginine in humans. Am J Physiol. 1995 Nov;269(5 Pt 1):E884-96. doi: 10.1152/ajpendo.1995.269.5.E884. PMID 7491940
- [Background] Berkowitz DE, White R, Li D, Minhas KM, Cernetich A, Kim S, Burke S, Shoukas AA, Nyhan D, Champion HC, Hare JM. Arginase reciprocally regulates nitric oxide synthase activity and contributes to endothelial dysfunction in aging blood vessels. Circulation. 2003 Oct 21;108(16):2000-6. doi: 10.1161/01.CIR.0000092948.04444.C7. Epub 2003 Sep 29. PMID 14517171
- [Background] Blackburn P, Lemieux I, Almeras N, Bergeron J, Cote M, Tremblay A, Lamarche B, Despres JP. The hypertriglyceridemic waist phenotype versus the National Cholesterol Education Program-Adult Treatment Panel III and International Diabetes Federation clinical criteria to identify high-risk men with an altered cardiometabolic risk profile. Metabolism. 2009 Aug;58(8):1123-30. doi: 10.1016/j.metabol.2009.03.012. Epub 2009 Jun 18. PMID 19481769
- [Background] Blackburn P, Lemieux I, Lamarche B, Bergeron J, Perron P, Tremblay G, Gaudet D, Despres JP. Hypertriglyceridemic waist: a simple clinical phenotype associated with coronary artery disease in women. Metabolism. 2012 Jan;61(1):56-64. doi: 10.1016/j.metabol.2011.05.017. Epub 2011 Jul 5. PMID 21733531
- [Background] Blum A, Hathaway L, Mincemoyer R, Schenke WH, Kirby M, Csako G, Waclawiw MA, Panza JA, Cannon RO 3rd. Effects of oral L-arginine on endothelium-dependent vasodilation and markers of inflammation in healthy postmenopausal women. J Am Coll Cardiol. 2000 Feb;35(2):271-6. doi: 10.1016/s0735-1097(99)00553-7. PMID 10676669
- [Background] Bode-Boger SM, Boger RH, Galland A, Tsikas D, Frolich JC. L-arginine-induced vasodilation in healthy humans: pharmacokinetic-pharmacodynamic relationship. Br J Clin Pharmacol. 1998 Nov;46(5):489-97. doi: 10.1046/j.1365-2125.1998.00803.x. PMID 9833603
- [Background] Bode-Boger SM, Muke J, Surdacki A, Brabant G, Boger RH, Frolich JC. Oral L-arginine improves endothelial function in healthy individuals older than 70 years. Vasc Med. 2003 May;8(2):77-81. doi: 10.1191/1358863x03vm474oa. PMID 14518608
- [Background] Bode-Boger SM. Effect of L-arginine supplementation on NO production in man. Eur J Clin Pharmacol. 2006;62:91-9
- [Background] Boger GI, Rudolph TK, Maas R, Schwedhelm E, Dumbadze E, Bierend A, Benndorf RA, Boger RH. Asymmetric dimethylarginine determines the improvement of endothelium-dependent vasodilation by simvastatin: Effect of combination with oral L-arginine. J Am Coll Cardiol. 2007 Jun 12;49(23):2274-82. doi: 10.1016/j.jacc.2007.02.051. Epub 2007 May 25. PMID 17560293
- [Background] Boger RH. The pharmacodynamics of L-arginine. J Nutr. 2007 Jun;137(6 Suppl 2):1650S-1655S. doi: 10.1093/jn/137.6.1650S. PMID 17513442
- [Background] Brunner H, Cockcroft JR, Deanfield J, Donald A, Ferrannini E, Halcox J, Kiowski W, Luscher TF, Mancia G, Natali A, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Spieker LE, Taddei S, Webb DJ; Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part II: Association with cardiovascular risk factors and diseases. A statement by the Working Group on Endothelins and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Feb;23(2):233-46. doi: 10.1097/00004872-200502000-00001. PMID 15662207
- [Background] Castillo L, Chapman TE, Yu YM, Ajami A, Burke JF, Young VR. Dietary arginine uptake by the splanchnic region in adult humans. Am J Physiol. 1993 Oct;265(4 Pt 1):E532-9. doi: 10.1152/ajpendo.1993.265.4.E532. PMID 8238326
- [Background] Castillo L, deRojas TC, Chapman TE, Vogt J, Burke JF, Tannenbaum SR, Young VR. Splanchnic metabolism of dietary arginine in relation to nitric oxide synthesis in normal adult man. Proc Natl Acad Sci U S A. 1993 Jan 1;90(1):193-7. doi: 10.1073/pnas.90.1.193. PMID 8419922
- [Background] Chan NN, Colhoun HM, Vallance P. Cardiovascular risk factors as determinants of endothelium-dependent and endothelium-independent vascular reactivity in the general population. J Am Coll Cardiol. 2001 Dec;38(7):1814-20. doi: 10.1016/s0735-1097(01)01669-2. PMID 11738279
- [Background] Deanfield J, Donald A, Ferri C, Giannattasio C, Halcox J, Halligan S, Lerman A, Mancia G, Oliver JJ, Pessina AC, Rizzoni D, Rossi GP, Salvetti A, Schiffrin EL, Taddei S, Webb DJ; Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. Endothelial function and dysfunction. Part I: Methodological issues for assessment in the different vascular beds: a statement by the Working Group on Endothelin and Endothelial Factors of the European Society of Hypertension. J Hypertens. 2005 Jan;23(1):7-17. doi: 10.1097/00004872-200501000-00004. PMID 15643116
- [Background] Despres JP, Lemieux I, Bergeron J, Pibarot P, Mathieu P, Larose E, Rodes-Cabau J, Bertrand OF, Poirier P. Abdominal obesity and the metabolic syndrome: contribution to global cardiometabolic risk. Arterioscler Thromb Vasc Biol. 2008 Jun;28(6):1039-49. doi: 10.1161/ATVBAHA.107.159228. Epub 2008 Mar 20. PMID 18356555
- [Background] Donald AE, Charakida M, Cole TJ, Friberg P, Chowienczyk PJ, Millasseau SC, Deanfield JE, Halcox JP. Non-invasive assessment of endothelial function: which technique? J Am Coll Cardiol. 2006 Nov 7;48(9):1846-50. doi: 10.1016/j.jacc.2006.07.039. Epub 2006 Oct 17. PMID 17084260
- [Background] Flammer AJ, Anderson T, Celermajer DS, Creager MA, Deanfield J, Ganz P, Hamburg NM, Luscher TF, Shechter M, Taddei S, Vita JA, Lerman A. The assessment of endothelial function: from research into clinical practice. Circulation. 2012 Aug 7;126(6):753-67. doi: 10.1161/CIRCULATIONAHA.112.093245. PMID 22869857
- [Background] Fouillet H, Juillet B, Gaudichon C, Mariotti F, Tome D, Bos C. Absorption kinetics are a key factor regulating postprandial protein metabolism in response to qualitative and quantitative variations in protein intake. Am J Physiol Regul Integr Comp Physiol. 2009 Dec;297(6):R1691-705. doi: 10.1152/ajpregu.00281.2009. Epub 2009 Oct 7. PMID 19812354
- [Background] Gomes VA, Casella-Filho A, Chagas AC, Tanus-Santos JE. Enhanced concentrations of relevant markers of nitric oxide formation after exercise training in patients with metabolic syndrome. Nitric Oxide. 2008 Dec;19(4):345-50. doi: 10.1016/j.niox.2008.08.005. Epub 2008 Sep 5. PMID 18799138
- [Background] Gomez-Huelgas R, Bernal-Lopez MR, Villalobos A, Mancera-Romero J, Baca-Osorio AJ, Jansen S, Guijarro R, Salgado F, Tinahones FJ, Serrano-Rios M. Hypertriglyceridemic waist: an alternative to the metabolic syndrome? Results of the IMAP Study (multidisciplinary intervention in primary care). Int J Obes (Lond). 2011 Feb;35(2):292-9. doi: 10.1038/ijo.2010.127. Epub 2010 Jun 15. PMID 20548300
- [Background] Grundy SM, Brewer HB Jr, Cleeman JI, Smith SC Jr, Lenfant C; National Heart, Lung, and Blood Institute; American Heart Association. Definition of metabolic syndrome: report of the National Heart, Lung, and Blood Institute/American Heart Association conference on scientific issues related to definition. Arterioscler Thromb Vasc Biol. 2004 Feb;24(2):e13-8. doi: 10.1161/01.ATV.0000111245.75752.C6. No abstract available. PMID 14766739
- [Background] Hill BG, Dranka BP, Bailey SM, Lancaster JR Jr, Darley-Usmar VM. What part of NO don't you understand? Some answers to the cardinal questions in nitric oxide biology. J Biol Chem. 2010 Jun 25;285(26):19699-704. doi: 10.1074/jbc.R110.101618. Epub 2010 Apr 21. PMID 20410298
- [Background] Joshi MS, Ferguson TB Jr, Johnson FK, Johnson RA, Parthasarathy S, Lancaster JR Jr. Receptor-mediated activation of nitric oxide synthesis by arginine in endothelial cells. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):9982-7. doi: 10.1073/pnas.0506824104. Epub 2007 May 29. PMID 17535904
- [Background] Kim JA, Montagnani M, Koh KK, Quon MJ. Reciprocal relationships between insulin resistance and endothelial dysfunction: molecular and pathophysiological mechanisms. Circulation. 2006 Apr 18;113(15):1888-904. doi: 10.1161/CIRCULATIONAHA.105.563213. PMID 16618833
- [Background] Lauer T, Heiss C, Balzer J, Kehmeier E, Mangold S, Leyendecker T, Rottler J, Meyer C, Merx MW, Kelm M, Rassaf T. Age-dependent endothelial dysfunction is associated with failure to increase plasma nitrite in response to exercise. Basic Res Cardiol. 2008 May;103(3):291-7. doi: 10.1007/s00395-008-0714-3. Epub 2008 Mar 17. PMID 18347836
- [Background] Li H, Forstermann U. Prevention of atherosclerosis by interference with the vascular nitric oxide system. Curr Pharm Des. 2009;15(27):3133-45. doi: 10.2174/138161209789058002. PMID 19754387
- [Background] Li Z, Wong A, Henning SM, Zhang Y, Jones A, Zerlin A, Thames G, Bowerman S, Tseng CH, Heber D. Hass avocado modulates postprandial vascular reactivity and postprandial inflammatory responses to a hamburger meal in healthy volunteers. Food Funct. 2013 Feb 26;4(3):384-91. doi: 10.1039/c2fo30226h. PMID 23196671
- [Background] Loscalzo J. What we know and don't know about L-arginine and NO. Circulation. 2000 May 9;101(18):2126-9. doi: 10.1161/01.cir.101.18.2126. No abstract available. PMID 10801749
- [Background] Luiking YC, Engelen MP, Deutz NE. Regulation of nitric oxide production in health and disease. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):97-104. doi: 10.1097/MCO.0b013e328332f99d. PMID 19841582
- [Background] Maas R, Schwedhelm E, Kahl L, Li H, Benndorf R, Luneburg N, Forstermann U, Boger RH. Simultaneous assessment of endothelial function, nitric oxide synthase activity, nitric oxide-mediated signaling, and oxidative stress in individuals with and without hypercholesterolemia. Clin Chem. 2008 Feb;54(2):292-300. doi: 10.1373/clinchem.2007.093575. Epub 2007 Dec 10. PMID 18070819
- [Background] Mariotti F, Huneau JF, Szezepanski I, Petzke KJ, Aggoun Y, Tome D, Bonnet D. Meal amino acids with varied levels of arginine do not affect postprandial vascular endothelial function in healthy young men. J Nutr. 2007 Jun;137(6):1383-9. doi: 10.1093/jn/137.6.1383. PMID 17513395
- [Background] Mariotti F, Mahe S, Luengo C, Benamouzig R, Tome D. Postprandial modulation of dietary and whole-body nitrogen utilization by carbohydrates in humans. Am J Clin Nutr. 2000 Oct;72(4):954-62. doi: 10.1093/ajcn/72.4.954. PMID 11010937
- [Background] Mariotti F, Petzke KJ, Bonnet D, Szezepanski I, Bos C, Huneau JF, Fouillet H. Kinetics of the utilization of dietary arginine for nitric oxide and urea synthesis: insight into the arginine-nitric oxide metabolic system in humans. Am J Clin Nutr. 2013 May;97(5):972-9. doi: 10.3945/ajcn.112.048025. Epub 2013 Mar 27. PMID 23535108
- [Background] Maxwell AJ. Mechanisms of dysfunction of the nitric oxide pathway in vascular diseases. Nitric Oxide. 2002 Mar;6(2):101-24. doi: 10.1006/niox.2001.0394. PMID 11890735
- [Background] McCrea CE, Skulas-Ray AC, Chow M, West SG. Test-retest reliability of pulse amplitude tonometry measures of vascular endothelial function: implications for clinical trial design. Vasc Med. 2012 Feb;17(1):29-36. doi: 10.1177/1358863X11433188. PMID 22363016
- [Background] Moncada S, Higgs EA. Molecular mechanisms and therapeutic strategies related to nitric oxide. FASEB J. 1995 Oct;9(13):1319-30. PMID 7557022
- [Background] Moncada S, Higgs EA. The discovery of nitric oxide and its role in vascular biology. Br J Pharmacol. 2006 Jan;147 Suppl 1(Suppl 1):S193-201. doi: 10.1038/sj.bjp.0706458. PMID 16402104
- [Background] Morris SM Jr. Recent advances in arginine metabolism: roles and regulation of the arginases. Br J Pharmacol. 2009 Jul;157(6):922-30. doi: 10.1111/j.1476-5381.2009.00278.x. Epub 2009 Jun 5. PMID 19508396
- [Background] Napoli C, de Nigris F, Williams-Ignarro S, Pignalosa O, Sica V, Ignarro LJ. Nitric oxide and atherosclerosis: an update. Nitric Oxide. 2006 Dec;15(4):265-79. doi: 10.1016/j.niox.2006.03.011. Epub 2006 Apr 15. PMID 16684613
- [Background] Nawabzad R, Champin B. [Concordance between three definitions for metabolic syndrome (Hypertriglyceridemic waist, National Cholesterol Education Program, International Diabetes Federation), and prevalence of the syndrome in a French population]. Rev Prat. 2010 Dec 20;60(10 Suppl):15-23. French. PMID 22530271
- [Background] Ohta F, Takagi T, Sato H, Ignarro LJ. Low-dose L-arginine administration increases microperfusion of hindlimb muscle without affecting blood pressure in rats. Proc Natl Acad Sci U S A. 2007 Jan 23;104(4):1407-11. doi: 10.1073/pnas.0610207104. Epub 2007 Jan 17. PMID 17229841
- [Background] Pfeuffer M, Fielitz K, Laue C, Winkler P, Rubin D, Helwig U, Giller K, Kammann J, Schwedhelm E, Boger RH, Bub A, Bell D, Schrezenmeir J. CLA does not impair endothelial function and decreases body weight as compared with safflower oil in overweight and obese male subjects. J Am Coll Nutr. 2011 Feb;30(1):19-28. doi: 10.1080/07315724.2011.10719940. PMID 21697535
- [Background] Preli RB, Klein KP, Herrington DM. Vascular effects of dietary L-arginine supplementation. Atherosclerosis. 2002 May;162(1):1-15. doi: 10.1016/s0021-9150(01)00717-1. PMID 11947892
- [Background] Rizzo NO, Maloney E, Pham M, Luttrell I, Wessells H, Tateya S, Daum G, Handa P, Schwartz MW, Kim F. Reduced NO-cGMP signaling contributes to vascular inflammation and insulin resistance induced by high-fat feeding. Arterioscler Thromb Vasc Biol. 2010 Apr;30(4):758-65. doi: 10.1161/ATVBAHA.109.199893. Epub 2010 Jan 21. PMID 20093624
- [Background] Schafer A, Wiesmann F, Neubauer S, Eigenthaler M, Bauersachs J, Channon KM. Rapid regulation of platelet activation in vivo by nitric oxide. Circulation. 2004 Apr 20;109(15):1819-22. doi: 10.1161/01.CIR.0000126837.88743.DD. Epub 2004 Apr 5. PMID 15066953
- [Background] Schwedhelm E, Maas R, Freese R, Jung D, Lukacs Z, Jambrecina A, Spickler W, Schulze F, Boger RH. Pharmacokinetic and pharmacodynamic properties of oral L-citrulline and L-arginine: impact on nitric oxide metabolism. Br J Clin Pharmacol. 2008 Jan;65(1):51-9. doi: 10.1111/j.1365-2125.2007.02990.x. Epub 2007 Jul 27. PMID 17662090
- [Background] Siani A, Pagano E, Iacone R, Iacoviello L, Scopacasa F, Strazzullo P. Blood pressure and metabolic changes during dietary L-arginine supplementation in humans. Am J Hypertens. 2000 May;13(5 Pt 1):547-51. doi: 10.1016/s0895-7061(99)00233-2. PMID 10826408
- [Background] Siekmeier R, Grammer T, Marz W. Roles of oxidants, nitric oxide, and asymmetric dimethylarginine in endothelial function. J Cardiovasc Pharmacol Ther. 2008 Dec;13(4):279-97. doi: 10.1177/1074248408326488. Epub 2008 Oct 22. PMID 18945874
- [Background] Siervo M, Jackson SJ, Bluck LJ. In-vivo nitric oxide synthesis is reduced in obese patients with metabolic syndrome: application of a novel stable isotopic method. J Hypertens. 2011 Aug;29(8):1515-27. doi: 10.1097/HJH.0b013e3283487806. PMID 21720276
- [Background] Siervo M, Stephan BC, Feelisch M, Bluck LJ. Measurement of in vivo nitric oxide synthesis in humans using stable isotopic methods: a systematic review. Free Radic Biol Med. 2011 Aug 15;51(4):795-804. doi: 10.1016/j.freeradbiomed.2011.05.032. Epub 2011 Jun 13. PMID 21672626
- [Background] Tangphao O, Grossmann M, Chalon S, Hoffman BB, Blaschke TF. Pharmacokinetics of intravenous and oral L-arginine in normal volunteers. Br J Clin Pharmacol. 1999 Mar;47(3):261-6. doi: 10.1046/j.1365-2125.1999.00883.x. PMID 10215749
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Background] Tousoulis D, Kampoli AM, Tentolouris C, Papageorgiou N, Stefanadis C. The role of nitric oxide on endothelial function. Curr Vasc Pharmacol. 2012 Jan;10(1):4-18. doi: 10.2174/157016112798829760. PMID 22112350
- [Background] Tsikas D, Boger RH, Sandmann J, Bode-Boger SM, Frolich JC. Endogenous nitric oxide synthase inhibitors are responsible for the L-arginine paradox. FEBS Lett. 2000 Jul 28;478(1-2):1-3. doi: 10.1016/s0014-5793(00)01686-0. PMID 10922458
- [Background] Voetsch B, Jin RC, Loscalzo J. Nitric oxide insufficiency and atherothrombosis. Histochem Cell Biol. 2004 Oct;122(4):353-67. doi: 10.1007/s00418-004-0675-z. Epub 2004 Aug 26. PMID 15338226
- [Background] Vogel RA, Corretti MC, Plotnick GD. Effect of a single high-fat meal on endothelial function in healthy subjects. Am J Cardiol. 1997 Feb 1;79(3):350-4. doi: 10.1016/s0002-9149(96)00760-6. PMID 9036757
- [Background] West SG, Likos-Krick A, Brown P, Mariotti F. Oral L-arginine improves hemodynamic responses to stress and reduces plasma homocysteine in hypercholesterolemic men. J Nutr. 2005 Feb;135(2):212-7. doi: 10.1093/jn/135.2.212. PMID 15671215
- [Background] Wilkinson IB, Qasem A, McEniery CM, Webb DJ, Avolio AP, Cockcroft JR. Nitric oxide regulates local arterial distensibility in vivo. Circulation. 2002 Jan 15;105(2):213-7. doi: 10.1161/hc0202.101970. PMID 11790703
- [Background] Wu G, Morris SM Jr. Arginine metabolism: nitric oxide and beyond. Biochem J. 1998 Nov 15;336 ( Pt 1)(Pt 1):1-17. doi: 10.1042/bj3360001. PMID 9806879
- [Background] Wu G, Meininger CJ. Arginine nutrition and cardiovascular function. J Nutr. 2000 Nov;130(11):2626-9. doi: 10.1093/jn/130.11.2626. PMID 11053497
- [Background] Wu G, Meininger CJ. Regulation of nitric oxide synthesis by dietary factors. Annu Rev Nutr. 2002;22:61-86. doi: 10.1146/annurev.nutr.22.110901.145329. Epub 2002 Jan 4. PMID 12055338
- [Background] Wyatt AW, Steinert JR, Mann GE. Modulation of the L-arginine/nitric oxide signalling pathway in vascular endothelial cells. Biochem Soc Symp. 2004;(71):143-56. doi: 10.1042/bss0710143. PMID 15777019
- [Background] Yang Z, Ming XF. Recent advances in understanding endothelial dysfunction in atherosclerosis. Clin Med Res. 2006 Mar;4(1):53-65. doi: 10.3121/cmr.4.1.53. PMID 16595793
- [Background] Skulas-Ray AC, Kris-Etherton PM, Harris WS, Vanden Heuvel JP, Wagner PR, West SG. Dose-response effects of omega-3 fatty acids on triglycerides, inflammation, and endothelial function in healthy persons with moderate hypertriglyceridemia. Am J Clin Nutr. 2011 Feb;93(2):243-52. doi: 10.3945/ajcn.110.003871. Epub 2010 Dec 15. PMID 21159789
- [Background] Hamburg NM, Benjamin EJ. Assessment of endothelial function using digital pulse amplitude tonometry. Trends Cardiovasc Med. 2009 Jan;19(1):6-11. doi: 10.1016/j.tcm.2009.03.001. PMID 19467447
- [Background] Herieka M, Erridge C. High-fat meal induced postprandial inflammation. Mol Nutr Food Res. 2014 Jan;58(1):136-46. doi: 10.1002/mnfr.201300104. Epub 2013 Jul 12. PMID 23847095
- [Derived] Dimina L, Tremblay-Franco M, Deveaux A, Tardivel C, Fouillet H, Polakof S, Martin JC, Mariotti F. Plasma Metabolome Analysis Suggests That L-Arginine Supplementation Affects Microbial Activity Resulting in a Decrease in Trimethylamine N-oxide-A Randomized Controlled Trial in Healthy Overweight Adults with Cardiometabolic Risk Factors. Curr Dev Nutr. 2023 Nov 20;7(12):102038. doi: 10.1016/j.cdnut.2023.102038. eCollection 2023 Dec. PMID 38162999
- [Derived] Deveaux A, Pham I, West SG, Andre E, Lantoine-Adam F, Bunouf P, Sadi S, Hermier D, Mathe V, Fouillet H, Huneau JF, Benamouzig R, Mariotti F. l-Arginine Supplementation Alleviates Postprandial Endothelial Dysfunction When Baseline Fasting Plasma Arginine Concentration Is Low: A Randomized Controlled Trial in Healthy Overweight Adults with Cardiometabolic Risk Factors. J Nutr. 2016 Jul;146(7):1330-40. doi: 10.3945/jn.115.227959. Epub 2016 Jun 8. PMID 27281800